CLINICAL TRIAL: NCT03818464
Title: Pre-operative Psychological Assessment of Patients Undergoing General Anesthesia in Abdominal Surgery
Brief Title: Psychological Assessment Before General Anesthesia (VeSPPA2018)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Elena Giovanna Bignami, Clinical Professor, University of Parma
Other Study IDs: 730/2018/OSS/AOUPR
Record Dates: First submitted 2019-01-21; First posted 2019-01-28 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia
Keywords: pre-operative assessment; postoperative pain; biological complications
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The level of preoperative anxiety can be related to the outcome of an operation and to the post operative patient management .

The Dutch questionnaire APAIS (Amsterdam Preoperative Anxiety and Information Scale) is a useful tool to quantify this parameter, and it has been translated and validated by the University Federico II of Naples in the study "Italian validation of the Amsterdam Preoperative Anxiety and Information Scale".

The study aims at identifying the correlation between the preoperative anxiety level measured by the APAIS in adult patients in general anesthesia undergoing elective major abdominal surgery and the levels of post-operative pain measured by the VAS (Visual Analogue Scale) and NRS (Numeric Rating Scale) scales.

Post-operative pain and agitation in the patient can be lessened through the objective assessment of preoperative anxiety and its treatment.

DETAILED DESCRIPTION:
Background and aim:

Anxiety is the body's physiological response to danger. It is a complex combination of emotions and fear, which leads to developing the typical symptoms of the "fight or flight" mode, as well as hyperactivity of the sympathetic nervous system which causes the body to release the adrenal "stress hormones" (cortisol, noradrenaline and adrenaline).

Anxiety reaction is commonly experienced by patients undergoing surgeries, as these are perceived as dangerous situations that cause the patient to feel powerless. Clinical practice has shown that patients are concerned not only about the surgery itself but also about the state of unconsciousness in which they enter because of general anesthesia. General anesthesia is a medically induced coma which is temporary and reversible. It is obtained by administering drugs to the patient, and it consists of three components - hypnosis, analgesia and muscle relaxation.

The procedure can be broken down in the following phases:

medication - the patient is administered anxiolytic drugs.

Induction of general anesthesia - loss of consciousness and respiratory arrest; breathing supported by mechanical ventilation.

Maintenance - surgery is carried out.

Emergence from anesthesia - administration of anesthetics is ceased and spontaneous breathing resumes.

Anxious patients have hyperarousal of the sympathetic nervous system, which affects the management of general anesthesia; with these patients, medication dosing will need to be adjusted in order to counterbalance the hemodynamic and metabolic consequences caused by this hyperarousal.

The following hypothesis is the aim of the study: to identify a significant number of correlations between the preoperative anxiety levels (quantified by the APAIS questionnaire), postoperative pain (quantified by the VAS and NRS scales), and the objective biological parameters displayed in the crf.

Gathering such data precedes considering whether the modulation of preoperative anxiety can affect positively the patient's outcome.

As a matter of fact, it is considered that reducing preoperative anxiety (for example through doctor-patient conversation or administration of anxiolytic drugs) allows an improving of postoperative physical and psychological conditions.

Medical literature on this topic shows that the preoperative anxiety level can be related to the outcome of an operation and to the post-operative patient management. In 1996, the Dutch Nelly Moerman, Martin J. Muller, F. S. van Dam and Hans Oosting introduced the Amsterdam Preoperative Anxiety and Information Scale (APAIS) - a scale for the objective assessment of anxiety.

It is a quick questionnaire consisting of 6 questions; its purpose is to investigate in detail the patient's anxiety and his/her need of information about general anesthesia and the surgery he/she will undergo. The questionnaire is easy to use and precise, which led to a widespread use of the APAIS scale.

In Italy, the APAIS scale has been the subject matter of the study "Italian validation of the Amsterdam Preoperative Anxiety and Information Scale" carried out by the the University Federico II of Naples. This study demonstrated that the scale measured effectively the preoperative anxiety level in that portion of Italian population undergoing surgery, and it reliably identifies pathological anxiety. In fact, there are cases in which anxiety is not an adaptive (thus physiological) response, but it reveals to be maladaptive (and thus pathological). When present in the preoperative phase, this type of anxiety can strongly affect a surgery's outcome.

The study aims at using the APAIS scale to measure preoperative anxiety levels in adult patients in general anesthesia undergoing elective major abdominal surgery, and then assess the correlation between the anxiety levels and the patient's wellbeing in the postoperative phase. The investigators believes that the management of both surgery and patient's postoperative pain can be improved through an objective assessment of preoperative anxiety and its treatment. The questionnaire allows to obtain a certain score corresponding to a certain level of anxiety in the patient (in the Italian translation of APAIS, the score >14 corresponds to "pathological anxiety"). The work aims at identifying a significant number of correlations between this score and the pain and between anxiety and the variation of biological parameters displayed in the cfr (frequency, blood pressure, hemoglobin, and so on).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged between 18 and 75 years.
* Degrees I, II and III of the ASA Classification (Classification of the physical condition of the patient).
* Patients under general anesthesia for major abdominal surgery in election.
* Adult aware and informed that he has signed the informed consent form.

Exclusion Criteria:

* Patient who refuses to sign informed consent.
* Patient under general anesthesia for emergency surgery.
* Patient with an established diagnosis and / or in therapy for serious diseases of the emotional sphere, major depression or severe psychosis.
* Patient with history of drug addiction and / or alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-critically ill patients undergoing general anesthesia before elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-10 (Estimated); Primary Completion 2020-02-10 (Estimated); Study Completion 2021-03-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between anxiety level and postoperative pain | from before induction of general anesthesia until the end of recovery, up to 3 days
  Identify the correlation between the preoperative patient anxiety level measured by APAIS (Amsterdam Preoperative Anxiety and Information Scale) and the postoperative pain levels measured using the VAS (Visual Analogue Scale). The evaluation range of Apais scale is from one (the lower level with better outcome) to five (the maximum level with worse outcome). The VAS Scale is made of six smiles from zero (the lower level with better outcome) to five ( the maximum level of pain with worse outcome).
Correlation between anxiety level and postoperative pain | from before induction of general anesthesia until the end of recovery, up to 3 days
  Identify the correlation between the preoperative patient anxiety level measured by APAIS (Amsterdam Preoperative Anxiety and Information Scale) and the postoperative pain levels measured using the NRS (Numeric Rating Scales). The evaluation range of Apais scale is from one (the lower level with better outcome) to five (the maximum level with worse outcome). The evaluation range of NRS scale is from zero ( the lower level with better outcome) to ten (the maximum level with worse outcome).
Level of agitation at the time of extubation | from the time of extubation until the end of recovery, up to 3 days
  Evaluate the level of agitation at the time of extubation through the BARS scale (Behavioral Activity Rating Scale). The evaluation range of the Bars scale is from one (the lower level with better outcome) to seven (the maximum level with worse outcome)
Level of agitation at the time of extubation | from the time of extubation until the end of recovery, up to 3 days
  Evaluate the level of agitation at the time of extubation through the RAMSAY Score (Ramsay Sedation Scale). The evaluation range of the Ramsay score is from one (the lower level with better outcome ) to six (the maximum level with worse outcome).

SECONDARY OUTCOMES:
Evaluate treatment of anxiety | from the time of awakening until the end of recovery, up to 3 days
  Pre-operative anxiety will be evaluated through APAIS (Amsterdam Preoperative Anxiety and Information Scale) questionnaire, for set the optimal type and dosage (mg/Kg) of drugs given for anxiety treatment.
Evaluate treatment of pain | from the time of awakening until the end of recovery, up to 3 days
  Post operative pain will be evaluated through VAS (Visual Analogue Scale) score, for set the optimal type and dosage (mg/Kg) of drugs given for pain treatment.
  The VAS Scale is made of six smiles from zero (the lower level with better outcome) to five ( the maximum level of pain with worse outcome).
Evaluate treatment of pain | from the time of awakening until the end of recovery, up to 3 days
  Post operative pain will be evaluated through NRS (Numeric Rating Scale) score, for set the optimal type and dosage (mg/Kg) of drugs given for pain treatment. The evaluation range of NRS scale is from zero ( the lower level with better outcome) to ten (the maximum level with worse outcome).
Patient's emotional background | from the time of awakening until the end of recovery, up to 3 days
  To investigate the patient's emotional background on the experience of general anesthesia through post-operative interviews
Neoplastic patient | from the time of awakening until the end of recovery, up to 3 days
  Evaluate the presence of any APAIS (Amsterdam Preoperative Anxiety and Information Scale) score differences in patients with and without neoplasia. The evaluation range of Apais scale is from one (the lower level with better outcome) to five (the maximum level with worse outcome)
Postoperative complications | from the time of awakening until the end of recovery, up to 3 days
  Evaluate the incidence of postoperative complications such as hypoxia, correlating the APAIS (Amsterdam Preoperative Anxiety and Information Scale) score in the preoperative with the values of arterial pressure, heart rate, oxygen saturation, hemoglobin and hematocrit in the postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella Troglio, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Andrea Bonetti, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Mirko Bottari, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Federica Cassè, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Federica Causo, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Jessica Colla, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; PierCarlo Cottone, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Marco DiLecce, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Giovanni Gasbarro, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Gelinda Giadone, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Valentina Giampaoli, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Filippo Grandini, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Vera Gualeni, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Alberto Iori, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Marcello LaBombarda, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Cristina Madoni, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Benedetta Marziani, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Cristina Piccinini, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- Azienda Ospedaliero-Universitaria di Parma, Parma, Italy (pr), Italy